CLINICAL TRIAL: NCT00597506
Title: Expanded Cohort of Patients With Refractory Metastatic Colorectal Cancer (MCRC) Treated With Bevacizumab and Everolimus
Brief Title: Expanded Cohort for Metastatic Colorectal Cancer (MCRC) Using Bevacizumab + Everolimus
Acronym: BEV/EV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herbert Hurwitz (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Herbert Hurwitz, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00001574
Record Dates: First submitted 2007-12-26; First posted 2008-01-18 (Estimated); Results first posted 2012-08-16 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: Colorectal Adenocarcinoma
Keywords: colorectal; refractory; adenocarcinoma; bevacizumab; everolimus
MeSH Terms: conditions — Adenocarcinoma | interventions — Bevacizumab; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab and Everolimus (Experimental): 10 mg Everolimus(RAD001) daily by mouth, days 1-28 10 mg/kg intravenous bevacizumab given days 1 and 15 of each cycle
  Interventions: Drug: Bevacizumab; Drug: Everolimus

INTERVENTIONS:
Drug: Bevacizumab — 10 mg/kg intravenous bevacizumab given days 1 and 15 of each cycle
  Other Names: Avastin
Drug: Everolimus — 10 mg Everolimus(RAD001) daily by mouth, days 1-28
  Other Names: RAD001

SUMMARY:
The purpose of this study is to find the safest and most effective dose of the drugs bevacizumab and everolimus given in combination for the treatment of metastatic colorectal cancer. Bevacizumab (also called Avastin™) is a drug that is given intravenously (through a vein). Everolimus (also called RAD001) is a tablet that is taken by mouth.

Bevacizumab is a protein that is thought to prevent the formation of blood vessels tumors need to grow. RAD001 has multiple capabilities, like bevacizumab it may prevent the formation of blood vessels needed by tumors and it also may stop tumor growth.

This study will try to find the safest dose of these drugs that can be tolerated when taken in combination. The study will look at how the drugs work in the body, and will see if there is any effect on metastatic colorectal cancer.

DETAILED DESCRIPTION:
This open-label, non-randomized expanded cohort trial of bevacizumab and RAD001 for patients with refractory metastatic colorectal cancer is designed to assess preliminary efficacy as well as the safety and tolerability of this combination. Patients will be accrued to this study at Duke University Medical Center and The Duke Oncology Outreach Network (DON)

After satisfying eligibility and screening criteria, patients will be treated on 28 day cycles.

* The treatment regimen is as follows:

  10 mg/kg Bevacizumab intravenous on days 1 and 15 and 10mg everolimus (RAD001) daily by mouth
* Toxicity will be assessed every visit, and as clinically indicated.
* Efficacy will be assessed every 2 cycles, and as clinically indicated.
* Patients may remain on treatment as long as they are deemed to be clinically benefiting from treatment, do not have progressive disease on restaging imaging (Section 6.0), or do not have any other reason for discontinuation of treatment as outlined in Section 3.4.
* Patients will undergo correlative studies as outlined in the study protocol

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed adenocarcinoma of the colon or rectum that has progressed on, or patient could not tolerate, fluoropyrimidine, oxaliplatin, irinotecan, and cetuximab and/or panitumumab chemotherapy. Disease must be measurable or evaluable by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Patients must not have had radiation therapy, hormonal therapy, biologic therapy or chemotherapy for cancer within the 28 days prior to study day 1. Patients must not have had major surgery within the 28 days prior to study day 1 or minor surgical procedures within the 7 days prior to study day 1.
* Age >18 years.
* Karnofsky performance status > 70 percent
* Life expectancy of at least 3 months.
* Patients must have normal organ and marrow function as defined in the protocol
* The effect of the investigational drugs on the developing human fetus is not known, but these drugs are likely to be embryo- and feto- toxic. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner are participating in this study, she should inform her treating physician and study PI immediately. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study. Patients who are pregnant and/or lactating are excluded from this study.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had radiation therapy, hormonal therapy, biologic therapy, or chemotherapy for cancer within the 28 days prior to day 1 of the study.
* Patients who have received any other investigational agents within the 28 days prior to day 1 of the study.
* Patients with known central nervous system (CNS) metastases.
* Inadequately controlled hypertension (defined as systolic blood pressure >150 and/or diastolic blood pressure > 100 mmHg). Initiation of antihypertensive is permitted provided adequate control is documented over at least 1 week before starting treatment.
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy. Patients on therapeutic anticoagulation may be enrolled provided that they have been clinically stable on anti-coagulation for at least 2 weeks.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment (56 days for hepatectomy, open thoracotomy, major neurosurgery) or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure excluding study-related procedures or placement of a vascular access device, within 7 days prior to expected start of treatment.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* Serious, non-healing wound, ulcer, or bone fracture
* Proteinuria at screening as demonstrated by either Urine protein:creatinine (UPC) ratio greater than or equal to 1.0 at screening
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix G)
* History of myocardial infarction, unstable angina, cardiac or other vascular stenting, angioplasty, or surgery within 6 months prior to study enrollment
* History of stroke or transient ischemic attack within 6 months prior to study enrollment
* History of intolerance or hypersensitivity to prior treatment with bevacizumab or RAD001.
* Chronic treatment with systemic steroids or another immunosuppressive agent, though steroids may be used on an as-needed basis - ie - for treatment of nausea. Treatment with megace or low dose glucocorticoids is permitted for treatment of anorexia.
* Other concurrent severe and/or uncontrolled medical disease which could compromise safety of treatment as so judged by treating physician
* A known history of HIV seropositivity, hepatitis C virus, acute or chronic active hepatitis B infection, or other serious chronic infection requiring ongoing treatment.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter drug absorption (e.g., inflammatory bowel disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or significant small bowel resection)
* Patients with an active, bleeding diathesis or on oral anti-vitamin K medication (except coumadin). No history of active GI bleeding or other major bleeding within previous 6 months.
* Patients unwilling to or unable to comply with the protocol
* Medical need for the continuous administration of any drugs which affect Cytochrome P450, family 3, subfamily A (CYP3A), though the use of low dose glucocorticoids for anorexia and /or nausea is permitted.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit safety or compliance with study requirements or may interfere with the interpretation of the results.
* History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or any evidence of interstitial lung disease on baseline chest CT scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert I Hurwitz, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment process started in October 2007 and was complete in April 2009. All subjects except one were enrolled at the Morris Cancer Clinic at Duke University Medical Center. One subject was enrolled at the Community Memorial Healthcenter in South Hill, Virgina which is a Duke Oncology Network clinical research site.
Groups:
- Drug: Bevacizumab and Everolimus: Open-label, non-randomized expanded cohort trial of refractory metastatic colorectal cancer subjects treated on 28 day cycles with the following treatment regimen: 10 mg/kg intravenous bevacizumab on days 1 and 15 each cycle and 10 mg everolimus(RAD001) daily by mouth.
Period: Overall Study
Arm/Group | Drug: Bevacizumab and Everolimus
Started | 50
Completed | 49
Not Completed | 1
Not completed — Subject is being followed for survival | 1

BASELINE CHARACTERISTICS:
Groups:
- Bevacizumab and Everolimus: Expanded Cohort of Patients with Refractory Metastatic Colorectal Cancer Treated With Bevacizumab and Everolimus
Arm/Group | Bevacizumab and Everolimus
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 56 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 30
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Overall Response
Description: Overall response is composed of complete responses and partial responses. Complete response (CR): disappearance of all target lesions; Partial response: at least a 30 percent decrease in the sum of the longest diameter of the target lesions taking as reference the baseline sum longest diameter. Response is assessed at each subject's restaging, approximately ever 2 months.
Time Frame: Measured 1 month after the last treated subject came off treatment
Population: 50 patients were enrolled and received bevacizumab at 10mg/kg every 2 weeks and everolimus at 10mg orally daily. However, only 49 patients were evaluable for progression. One patient who received less than 1 cycle of the regimen and died from a non-treatment-related illness was not included in the analysis.
Measure: Number; unit: percentage of participants
Groups:
- Bevacizumab and Everolimus: Enrolled participants on research study received bevacizumab at 10mg/kg every 2 weeks (day 1 and day 15 of each 28 day cycle) and everolimus at 10mg orally daily
Arm/Group | Bevacizumab and Everolimus
Number analyzed (Participants) | 49
percentage of participants | 0

2. Primary Outcome: Progression Free Survival (PFS)
Description: 8 week PFS
Time Frame: interval between start of treatment and 8-week
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Bevacizumab and Everolimus
Number analyzed (Participants) | 49
proportion of participants | 0.58 [0.46 to 0.68]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from 26Oct2007 (date of enrollment of first subject) through 17 April2010 (30 days after the last subject completed study drug).
Arm/Group | Bevacizumab and Everolimus
Serious Adverse Events (participants affected / at risk) | 27/50
Other Adverse Events (participants affected / at risk) | 48/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab and Everolimus (N=50)
Dehydration (Gastrointestinal disorders) | 2 (4)
Enterovesicular fistula (Gastrointestinal disorders) | 1 (1)
Bowel Perforation (Gastrointestinal disorders) | 1 (1)
Hemorrhage, GI rectum (Gastrointestinal disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Abdominal abscess with anastomatic leak (Gastrointestinal disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Infections and infestations) | 1 (1)
Pain (General disorders) | 1 (1)
Shortness of breath/chest pain (General disorders) | 1 (1)
Small bowel obstruction and pain (Gastrointestinal disorders) | 1 (1)
atrial fibrillation (Cardiac disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Cardiopulmonary arrest (Cardiac disorders) | 1 (1)
Abdominal pain (General disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aspiration (Gastrointestinal disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Disease progression/Death (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (2)
Acute Renal failure (Metabolism and nutrition disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab and Everolimus (N=50)
Hypokalemia (Metabolism and nutrition disorders) | 7
Hyperglycemia (Metabolism and nutrition disorders) | 6
Alkaline phosphatase elevation (Metabolism and nutrition disorders) | 6
Mucositis/Proctitis (Gastrointestinal disorders) | 37 — All grades of mucositis and proctitis
Hyperlipidemia (Metabolism and nutrition disorders) | 34
Hypertension (Cardiac disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes